CLINICAL TRIAL: NCT07236112
Title: A Prospective, Randomized, Open-label, Phase I Study of TRDC002 in the Diagnosis of Patients With PSMA-positive Recurrent or Metastatic Prostate Cancer
Brief Title: Study of TRDC002 in the Diagnosis of Patients With PSMA-positive Prostate Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: C Ray Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: TR1229
Record Dates: First submitted 2025-11-13; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; PSMA PET
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Enrolled participants will be randomized to receive a single dose of either 4 or 6 mCi of TRDC002.
Who Masked: Outcomes Assessor
Masking Description: Three independent readers will be blinded to all participants information and doses administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 4 mCi of TRDC002 (Experimental): Patients receive 4±0.5mCi (148±18.5 MBq) of TRDC002 IV. Patients then undergo PET/CT scan.
  Interventions: Drug: Intravenous (IV) single dose
- 6 mCi of TRDC002 (Experimental): Patients receive 6±0.5mCi (222±18.5 MBq) of TRDC002 IV. Patients then undergo PET/CT scan.
  Interventions: Drug: Intravenous (IV) single dose

INTERVENTIONS:
Drug: Intravenous (IV) single dose — Drug: TRDC002 A single dose of TRDC002 IV. Diagnostic Test: PET/CT imaging.

SUMMARY:
TRDC002 uses a radioactive form (64Cu) to trace the PSMA positive prostate cancer. The purpose of this study is to investigate TRDC002 as a PSMA PET tracer to localize PSMA positive lesions in adult patients with recurrent or metastatic prostate cancer. We plan to assess the PSMA PET/CT image quality following administration of two dose levels of TRDC002 to determine an acceptable dose and optimal acquisition time for obtaining diagnostic quality PET/CT images. The safety and tolerability, PK, biodistribution, dosimetry of TRDC002 will also be evaluated in this study.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label, phase I study to evaluate safety and tolerability, PK, biodistribution, dosimetry and preliminary efficacy of TRDC002 for PET/CT imaging in participants with PSMA-positive recurrent or metastatic prostate cancer compared with CRS.

At screening, the participants will be assessed for eligibility and will undergo PSMA PET to screen PSMA positive patients.

Eligible participants with recurrent or metastatic prostate cancer will be randomized to receive a single dose of either 4 or 6 mCi of TRDC002 intravenously. Whole-body PET/CT images will be acquired at 1hr, 4hr, 7hr, and 24hr post-injection to observe radiation absorbed dose and pharmacokinetics. Independent review committee (IRC) will evaluate the quality of PET images to determine an acceptable dose and optimal acquisition time for PET scan, and preliminary efficacy compared with Composite Reference Standard (CRS) based on CT/MRI with contrast and bone scan.

ELIGIBILITY:
Inclusion Criteria:

* Participants with recurrence or metastasis of prostate cancer.
* Participants with PSMA-positive lesions.
* Participants must have adequate bone marrow and organ function.
* Participants with an ECOG performance status of 0 or 1.

Exclusion Criteria:

* Any immunotherapy or biological therapy (including antibodies) targeting PSMA within 60 days prior to the day of randomization.
* A superscan is observed in the baseline bone scan.
* Concurrent serious (as determined by the Investigator) medical conditions
* Participants with symptomatic brain metastases, meningeal metastases, or spinal cord compression.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
the safety and tolerability of TRDC002 in participants | 3 days
  Adverse events (AEs) will be assessed and graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Pharmacokinetics of TRDC002. | Within 1 minute, 10 minutes, and 30 minutes, and at 60 minutes, 2 hours, 6 hours and 24 hours for blood PK, and 0-60 minutes, 1-2 hours, 2-6 hours, and 6-24 hours for urine PK.
  Peak plasma concentration (Cmax) will be performed by a bioanalytical HPLC method, free 64Cu, and known radiolysis byproducts of TRDC002 in plasma and urine samples.
Pharmacokinetics of TRDC002. | Within 1 minute, 10 minutes, and 30 minutes, and at 60 minutes, 2 hours, 6 hours and 24 hours for blood PK, and 0-60 minutes, 1-2 hours, 2-6 hours, and 6-24 hours for urine PK.
  Area under the plasma concentration versus time curve (AUC) will be performed by a bioanalytical HPLC method, free 64Cu, and known radiolysis byproducts of TRDC002 in plasma and urine samples.
Pharmacokinetics of TRDC002. | Within 1 minute, 10 minutes, and 30 minutes, and at 60 minutes, 2 hours, 6 hours and 24 hours for blood PK, and 0-60 minutes, 1-2 hours, 2-6 hours, and 6-24 hours for urine PK.
  Apparent elimination half-life (T1/2) will be performed by a bioanalytical HPLC method, free 64Cu, and known radiolysis byproducts of TRDC002 in plasma and urine samples.
The biodistribution of TRDC002. | At 1 hour, 4 hours, 7 hours, and 24 hours post injection.
  Biodistribution will be performed by average Standardized Uptake Value Maximum (SUVmax) of TRDC002 uptake in healthy organs and tumors.
The biodistribution of TRDC002. | At 1 hour, 4 hours, 7 hours, and 24 hours post injection.
  Biodistribution will be performed by average Standardized Uptake Value Mean (SUVmean) of TRDC002 uptake in healthy organs and tumors.
The biodistribution of TRDC002. | At 1 hour, 4 hours, 7 hours, and 24 hours post injection.
  Biodistribution will be performed by average injective dose (%ID) of TRDC002 uptake in healthy organs and tumors.
The dosimetry of TRDC002. | At 1 hour, 4 hours, 7 hours, and 24 hours post injection.
  Dosimetry will be assessed by absorbed dose.
The dosimetry of TRDC002. | At 1 hour, 4 hours, 7 hours, and 24 hours post injection.
  Dosimetry will be assessed by absorbed dose coefficients (ADC).
The dosimetry of TRDC002. | At 1 hour, 4 hours, 7 hours, and 24 hours post injection.
  Dosimetry will be assessed by effective dose.
The dosimetry of TRDC002. | At 1 hour, 4 hours, 7 hours, and 24 hours post injection.
  Dosimetry will be assessed by effective dose per administered activity.
The dosimetry of TRDC002. | At 1 hour, 4 hours, 7 hours, and 24 hours post injection.
  Dosimetry will be assessed by residence time.
PET/CT images to determine an acceptable dose and optimal acquisition time of PET scan. | At 1 hour, 4 hours, 7 hours, and 24 hours post injection.
  Image quality score will be used to judge the optimal dose level yielding diagnostic images at optimal acquisition time post-injection by majority of three readers.
PET/CT images to determine an acceptable dose and optimal acquisition time of PET scan. | At 1 hour, 4 hours, 7 hours, and 24 hours post injection.
  Signal-to-noise ratio (SNR) will be used to judge the optimal dose level yielding diagnostic images at optimal acquisition time post-injection by majority of three readers.
PET/CT images to determine an acceptable dose and optimal acquisition time of PET scan. | At 1 hour, 4 hours, 7 hours, and 24 hours post injection.
  Tumor-to-background ratio (TBR) will be used to judge the optimal dose level yielding diagnostic images at optimal acquisition time post-injection by majority of three readers.
PET/CT images to determine an acceptable dose and optimal acquisition time of PET scan. | At 1 hour, 4 hours, 7 hours, and 24 hours post injection.
  Lesion-to-blood pool ratio (LBR) will be used to judge the optimal dose level yielding diagnostic images at optimal acquisition time post-injection by majority of three readers.
PET/CT images to determine an acceptable dose and optimal acquisition time of PET scan. | At 1 hour, 4 hours, 7 hours, and 24 hours post injection.
  Lesion-to -muscle ratio (LMR) will be used to judge the optimal dose level yielding diagnostic images at optimal acquisition time post-injection by majority of three readers.

OTHER OUTCOMES:
The correct localization rate (CLR) of TRDC002 PET/CT imaging | At 1 hour, 4 hours, 7 hours, and 24 hours post injection.
  The region-level correct localization rate (CLR) of TRDC002 PET/CT imaging at different timepoints after administration.
The patient-level correct detection rate (CDR) of TRDC002 PET/CT imaging | At 1 hour, 4 hours, 7 hours, and 24 hours post injection.
  The patient-level correct detection rate (CDR) of TRDC002 PET/CT imaging for the detection of recurrent or metastatic prostate cancer at different timepoints after administration.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wu, MD, Study Chair — C Ray Therapeutics (Chengdu) Co., Ltd.
Locations (1):
- Union Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
We regret to inform you that we do not plan to share the Individual Participant Data (IPD) of this study due to the limited sample size. Thanks for your kind understanding.